CLINICAL TRIAL: NCT00012207
Title: A Phase I Study To Evaluate The Safety Of Cellular Immunotherapy Using Genetically Modified Autologous Cd20-Specific Cd8+ T Cell Clones For Patients With Relapsed Cd20+ Indolent Lymphomas
Brief Title: Biological Therapy After Chemotherapy in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1503.00; FHCRC-1503.00; NCI-G01-1921; CDR0000068494 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aldesleukin; Cyclophosphamide; Prednisone; Vincristine; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic autologous lymphocytes
Drug: cyclophosphamide
Drug: prednisone
Drug: vincristine sulfate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining biological therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of biological therapy after chemotherapy in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and toxicity of cellular immunotherapy with autologous CD8+ cytotoxic T-lymphocyte clones after chemotherapy comprising cyclophosphamide, vincristine, and prednisone in patients with relapsed or refractory CD20+ indolent lymphomas or mantle cell lymphoma.

Secondary

* Determine the duration of in vivo persistence of adoptively transferred CD20-specific CD8+ cytotoxic T-lymphocyte clones in the absence and presence of subcutaneous interleukin-2 in these patients.
* Assess the trafficking of CD8+ cytotoxic T-lymphocyte clones to lymph nodes in these patients treated with this regimen.
* Determine immune response and tumor response in patients treated with this regimen.

OUTLINE: This is an open-label, pilot study.

* Leukapheresis: Patients undergo leukapheresis. Selected CD20-specific CD8+ cells are cultured to expand the cytotoxic T lymphocytes (CTL), which are then cloned.
* Chemotherapy:

Patients receive oral cyclophosphamide and oral prednisone on days 1-5 and vincristine IV on day 1. Courses repeat every 3-4 weeks for a total of 6 courses.

* Immune cell infusion:

Beginning 4 weeks after the last course of chemotherapy (and lymph nodes ≤ 5 cm diameter or ≤ 5,000 circulating CD20+ lymphocytes/mm^3), patients receive autologous CD8+ CTL clones IV over 30 minutes. Courses repeat every 2-5 days for a total of 3 courses in the absence of disease progression or unacceptable toxicity. The last 6 patients receive interleukin-2 subcutaneously every 12 hours for 14 days, beginning 2 hours after the last infusion of CD8+ CTL clones.

After course 2 or 3 of immune cells, all patients undergo surgical lymph node biopsy to determine if immune cells are moving to the lymph nodes.

Patients are followed monthly for 1 year and then annually for 2 years.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Immunohistopathologically documented relapsed or refractory CD20+ indolent lymphomas or mantle cell lymphoma

  * Indolent B-cell lymphomas including any of the following subtypes:

    * Follicular lymphoma (grade I, II, or III)
    * Small lymphocytic lymphoma or chronic lymphocytic leukemia
    * Marginal zone lymphoma (splenic, nodal, and extra-nodal)
    * Lymphoplasmacytoid lymphoma
* Ineligible for or unwilling to participate in other FHCRC/UWMC protocols
* Serological evidence of prior exposure to Epstein-Barr virus
* Must agree to undergo peripheral blood drawing, bone marrow biopsy, lymph node biopsy, and nuclear medicine imaging
* Must agree to cytoreductive chemotherapy if necessary to reduce lymph nodes to < 5 cm in diameter or circulating B lymphocyte counts to < 5,000/mm^3
* No pulmonary involvement
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* At least 90 days

Hematopoietic:

* Not specified

Hepatic:

* No active hepatitis B infection

Renal:

* Not specified

Other:

* No HIV positivity
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of hypersensitivity reactions to murine proteins

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 months since prior rituximab, tositumomab, or ibritumomab
* No prior allogeneic stem cell transplantation
* No other concurrent immunotherapy (e.g., interferons, vaccines, or other cellular products)

Chemotherapy:

* At least 2 years since prior fludarabine or cladribine
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* No concurrent systemic corticosteroids except to treat toxicity from chemotherapy or cellular immunotherapy

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 4 weeks since prior immunosuppressive therapy and recovered
* No concurrent pentoxifylline
* No other concurrent investigational agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2000-09; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity by NCI CTC toxicity scale in patients w/ recurr. or refract. CD20+ follicular lymphoma who are not candidates for high dose chemoradiotx and stem cell transplant during each infusion, weekly for 4 wks and then monthly for a yr

SECONDARY OUTCOMES:
Duration of in vivo persistence of adoptively transferred CD20-specific CD8+ T cell clones by flow cytometry and quantitative polymerase chain reaction (qPCR) during each infusion, weekly for 4 weeks, and then monthly for a year
Trafficking of CD8+ CD20-specific T cell clones to lymph nodes by Gamma camera imaging during each infusion, weekly for 4 weeks, and then monthly for a year
Development of host anti-scFvFc:zeta (and anti-NeoR) immune responses by ELISA and chromium release assays during each infusion, weekly for 4 weeks, and then monthly for a year
Tumor responses to cyclophosphamide, vincristine, and prednisone (CVP) and to cytotoxic T-lymphocyte (CTL) infusions by Cheson criteria during each infusion, weekly for 4 weeks, and then monthly for a year

CONTACTS AND LOCATIONS:
Overall Officials: Oliver W. Press, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (3):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- [Result] Till BG, Jensen MC, Wang J, Chen EY, Wood BL, Greisman HA, Qian X, James SE, Raubitschek A, Forman SJ, Gopal AK, Pagel JM, Lindgren CG, Greenberg PD, Riddell SR, Press OW. Adoptive immunotherapy for indolent non-Hodgkin lymphoma and mantle cell lymphoma using genetically modified autologous CD20-specific T cells. Blood. 2008 Sep 15;112(6):2261-71. doi: 10.1182/blood-2007-12-128843. Epub 2008 May 28. PMID 18509084